CLINICAL TRIAL: NCT05047627
Title: Digital Intervention to Treat Anxiety and Depression Among Persons Receiving Treatment for Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, Nicholas Jacobson, Principal Investigator, Trustees of Dartmouth College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AWD00010555
Record Dates: First submitted 2021-08-13; First posted 2021-09-17 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Opioid-use Disorder; Anxiety Disorders; Depressive Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone Digital Intervention Group (Experimental): The Smartphone Digital Intervention Group is the experimental group. Participants randomized to this group will download the smartphone intervention and be asked to use the intervention four times per week for four weeks ( 16 digital sessions). The smartphone digital intervention will also continuously collect passive sensing data. The smartphone digital intervention will be designed to treat anxiety and depression by providing informational videos to help participants treat these symptoms. These videos include information about physical activity, muscle relaxation, and other proven helpful interventions to help with anxiety and depression.
  Interventions: Behavioral: Smartphone-Based Digital Intervention
- Wait list Control Condition (No Intervention): The wait list control condition will not receive the digital intervention treatment for the duration of the study. They will still provide urine samples during the study. Participants assigned to this condition will be able to access the digital intervention after their participation in the study.

INTERVENTIONS:
Behavioral: Smartphone-Based Digital Intervention — The digital intervention will be a prototype, and the current trial will be used to continue to both develop and refine the intervention. The current intervention will be based on a combination of cognitive-behavioral principles. As with prior research, the mobile platform will be delivered via Qualtrics, a HIPAA compliant and mobile-friendly platform. The cognitive-behavioral therapy will be primarily based on components with strongest support in digital interventions. The app will continuously collect passive sensing data on patterns in 1) sleep duration and quality;(2) light (3) location; (4) movement (5) social contact including duration and frequency of incoming and outcoming calls and text messages; (6) screen time; and (7) heart rate variability; (8) sound levels captured through passively collected smartphone The platform will deliver interactive interventions where participants will view texts and images, and it will also allow user interaction.
  Arms: Smartphone Digital Intervention Group

SUMMARY:
The majority of opioid users meet criteria for anxiety and depressive disorders, but most substance use disorder treatment programs do not offer treatment for co-occurring mental health problems. Anxiety and depression may also be directly linked to opioid use itself. Although treatments have been developed for anxiety and depressive symptoms for opioid users within face-to-face settings, few treatment facilities offer these in-person interventions due to their high cost and time burden. Given the deficits in research on treatments for anxiety and depression among those with opioid use disorder, the current research will examine the efficacy of a digital intervention designed to treat anxiety and depressive symptoms by augmenting the state of the science medication-based opioid use disorder treatment. Over the course of the proposed study, the research team will design and test the feasibility and acceptability of a standalone mobile intervention designed to treat persons receiving medication treatment for opioid use disorder. Participants receiving medication treatment for opioid use disorder will be randomized to receive a digital intervention to treat anxiety and depression or care as usual for a total of four weeks. The overarching goal of the proposed work is to test the feasibility and acceptability of the proposed mobile intervention. The Investigators will also explore the preliminary efficacy by examining reductions in anxiety and depressive symptoms and opioid cravings and use. This work could lead to a low-cost scalable solution to augment gold-standard treatment as usual in opioid use disorder by decreasing levels of comorbidity of anxiety and depressive disorders, thereby ultimately improving the outcomes of opioid use disorder itself.

DETAILED DESCRIPTION:
The study team will recruit a population of 60 adults who are receiving medication treatment for OUD from an online study based on Google Adwords, Reddit, and Facebook advertisements as online recruitment has been shown to be a viable and cost-effective recruitment method for opioid users. The total sample size may be expanded if recruitment costs are lower than expected.

Participants will complete self-report assessments on their anxiety symptoms, depressive symptoms, opioid cravings, and opioid use behaviors. Participants will be randomized to a smartphone-based digital intervention or waitlist control condition. The digital intervention will be designed to treat participants' anxiety and depressive symptoms, and participants will be asked to use the intervention four times per week for four weeks (16 digital sessions).The smartphone intervention will also collect passive sensing data continuously during the 4 week period. Participants will complete post measures and one-month follow-up measures on anxiety symptoms, depressive symptoms, opioid cravings, and opioid use behaviors. The urine drug screen will be mailed to participants. Participants will also be asked to complete five urine tests to detect substance use (amphetamines, barbiturates, benzodiazepines, cocaine, ecstasy, marijuana, methamphetamine, opioids, oxycodone, and pcp) across the study (1 at pre-digital intervention, 1 during the digital intervention, 1 post-digital intervention, 1 between post and follow-up of the digital intervention, and 1 at the 1-month follow-up of the digital intervention). Participants will be instructed when to complete each urine test and will be asked to take a photo of the back the label of each test showing the results to the experimenters and to text these photos to a Google Voice Number maintained by the experimenters.

Thus, this proposal seeks to address a crucial deficit in the availability of treatments for anxiety and depressive disorders among persons with OUD to ultimately augment treatment for OUD.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 or older)
* fluent in English
* able to provide informed consent
* meet current criteria for OUD (as defined by a Rapid Opioid Dependence Screen)
* are receiving methadone, buprenorphine, and/or naltrexone for OUD
* meet current criteria for an anxiety and/or depressive disorder (based on the Patient Health Questionnaire and the Generalized Anxiety Disorder Questionnaire).

Exclusion Criteria:

* active suicidality
* psychosis
* bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas C Jacobson, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Center For Technology and Behavioral Health, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Applebaum AJ, Bullis JR, Traeger LN, O'cleirigh C, Otto MW, Pollack MH, Safren SA. Rates of mood and anxiety disorders and contributors to continued heroin use in methadone maintenance patients: A comparison by HIV status. Neurobehav HIV Med. 2010 Aug 10;2010(2):49-57. doi: 10.2147/NBHIV.S12371. PMID 24062619
- [Background] Barry DT, Beitel M, Breuer T, Cutter CJ, Savant J, Peters S, Schottenfeld RS, Rounsaville BJ. Group-based strategies for stress reduction in methadone maintenance treatment: what do patients want? J Addict Med. 2011 Sep;5(3):181-7. doi: 10.1097/ADM.0b013e3181ee77cl. PMID 21841430
- [Background] Bartoli F, Carra G, Brambilla G, Carretta D, Crocamo C, Neufeind J, Baldacchino A, Humphris G, Clerici M. Association between depression and non-fatal overdoses among drug users: a systematic review and meta-analysis. Drug Alcohol Depend. 2014 Jan 1;134:12-21. doi: 10.1016/j.drugalcdep.2013.10.007. Epub 2013 Oct 24. PMID 24210424
- [Background] Blume, A. W., Schmaling, K. B., & Marlatt, G. A. (2000). Revisiting the self-medication hypothesis from a behavioral perspective. Cognitive and Behavioral Practice, 7(4), 379-384. https://doi.org/10.1016/S1077-7229(00)80048-6
- [Background] Borkovec TD, Newman MG, Pincus AL, Lytle R. A component analysis of cognitive-behavioral therapy for generalized anxiety disorder and the role of interpersonal problems. J Consult Clin Psychol. 2002 Apr;70(2):288-98. PMID 11952187
- [Background] Childress AR, Ehrman R, McLellan AT, MacRae J, Natale M, O'Brien CP. Can induced moods trigger drug-related responses in opiate abuse patients? J Subst Abuse Treat. 1994 Jan-Feb;11(1):17-23. doi: 10.1016/0740-5472(94)90060-4. PMID 8201629
- [Background] Cunningham JA, Hendershot CS, Kay-Lambkin F, Neighbors C, Griffiths KM, Bennett K, Bennett A, Godinho A, Schell C. Does providing a brief internet intervention for hazardous alcohol use to people seeking online help for depression reduce both alcohol use and depression symptoms among participants with these co-occurring disorders? Study protocol for a randomised controlled trial. BMJ Open. 2018 Jul 19;8(7):e022412. doi: 10.1136/bmjopen-2018-022412. PMID 30030322
- [Background] Deady M, Mills KL, Teesson M, Kay-Lambkin F. An Online Intervention for Co-Occurring Depression and Problematic Alcohol Use in Young People: Primary Outcomes From a Randomized Controlled Trial. J Med Internet Res. 2016 Mar 23;18(3):e71. doi: 10.2196/jmir.5178. PMID 27009465
- [Background] Firth J, Torous J, Nicholas J, Carney R, Pratap A, Rosenbaum S, Sarris J. The efficacy of smartphone-based mental health interventions for depressive symptoms: a meta-analysis of randomized controlled trials. World Psychiatry. 2017 Oct;16(3):287-298. doi: 10.1002/wps.20472. PMID 28941113
- [Background] Firth J, Torous J, Nicholas J, Carney R, Rosenbaum S, Sarris J. Can smartphone mental health interventions reduce symptoms of anxiety? A meta-analysis of randomized controlled trials. J Affect Disord. 2017 Aug 15;218:15-22. doi: 10.1016/j.jad.2017.04.046. Epub 2017 Apr 25. PMID 28456072
- [Background] Hassan AN, Howe AS, Samokhvalov AV, Le Foll B, George TP. Management of mood and anxiety disorders in patients receiving opioid agonist therapy: Review and meta-analysis. Am J Addict. 2017 Sep;26(6):551-563. doi: 10.1111/ajad.12581. Epub 2017 Jul 4. PMID 28675762
- [Background] Hogarth L, Hardy L, Bakou A, Mahlberg J, Weidemann G, Cashel S, Moustafa AA. Negative Mood Induction Increases Choice of Heroin Versus Food Pictures in Opiate-Dependent Individuals: Correlation With Self-Medication Coping Motives and Subjective Reactivity. Front Psychiatry. 2019 May 15;10:274. doi: 10.3389/fpsyt.2019.00274. eCollection 2019. PMID 31156470
- [Background] Hyman SM, Fox H, Hong KI, Doebrick C, Sinha R. Stress and drug-cue-induced craving in opioid-dependent individuals in naltrexone treatment. Exp Clin Psychopharmacol. 2007 Apr;15(2):134-43. doi: 10.1037/1064-1297.15.2.134. PMID 17469937
- [Background] Kay-Lambkin FJ, Baker AL, Lewin TJ, Carr VJ. Computer-based psychological treatment for comorbid depression and problematic alcohol and/or cannabis use: a randomized controlled trial of clinical efficacy. Addiction. 2009 Mar;104(3):378-88. doi: 10.1111/j.1360-0443.2008.02444.x. PMID 19207345
- [Background] Kenardy JA, Dow MG, Johnston DW, Newman MG, Thomson A, Taylor CB. A comparison of delivery methods of cognitive-behavioral therapy for panic disorder: an international multicenter trial. J Consult Clin Psychol. 2003 Dec;71(6):1068-75. doi: 10.1037/0022-006X.71.6.1068. PMID 14622082
- [Background] Kosten TR, Rounsaville BJ, Kleber HD. A 2.5-year follow-up of depression, life crises, and treatment effects on abstinence among opioid addicts. Arch Gen Psychiatry. 1986 Aug;43(8):733-8. doi: 10.1001/archpsyc.1986.01800080019003. PMID 3729667
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kroenke, Kurt, & Spitzer, R. L. (2002). The PHQ-9: A new depression diagnostic and severity measure. Psychiatric Annals, 32(9), 509-515. https://doi.org/10.3928/0048-5713-20020901-06
- [Background] Krupnick JL, Green BL, Amdur R, Alaoui A, Belouali A, Roberge E, Cueva D, Roberts M, Melnikoff E, Dutton MA. An Internet-based writing intervention for PTSD in veterans: A feasibility and pilot effectiveness trial. Psychol Trauma. 2017 Jul;9(4):461-470. doi: 10.1037/tra0000176. Epub 2016 Sep 8. PMID 27607767
- [Background] Lange A, Rietdijk D, Hudcovicova M, van de Ven JP, Schrieken B, Emmelkamp PM. Interapy: a controlled randomized trial of the standardized treatment of posttraumatic stress through the internet. J Consult Clin Psychol. 2003 Oct;71(5):901-9. doi: 10.1037/0022-006X.71.5.901. PMID 14516238
- [Background] Levin ME, Navarro C, Cruz RA, Haeger J. Comparing in-the-moment skill coaching effects from tailored versus non-tailored acceptance and commitment therapy mobile apps in a non-clinical sample. Cogn Behav Ther. 2019 May;48(3):200-216. doi: 10.1080/16506073.2018.1503706. Epub 2018 Aug 17. PMID 30117784
- [Background] Maloney E, Degenhardt L, Darke S, Nelson EC. Are non-fatal opioid overdoses misclassified suicide attempts? Comparing the associated correlates. Addict Behav. 2009 Sep;34(9):723-9. doi: 10.1016/j.addbeh.2009.04.011. Epub 2009 May 3. PMID 19447563
- [Background] Marshall BDL, Green TC, Elston B, Yedinak JL, Hadland SE, Clark MA. The Effectiveness of Internet- and Field-Based Methods to Recruit Young Adults Who Use Prescription Opioids Nonmedically. Subst Use Misuse. 2018 Aug 24;53(10):1688-1699. doi: 10.1080/10826084.2018.1425725. Epub 2018 Jan 24. PMID 29364768
- [Background] McHugh RK, Fitzmaurice GM, Carroll KM, Griffin ML, Hill KP, Wasan AD, Weiss RD. Assessing craving and its relationship to subsequent prescription opioid use among treatment-seeking prescription opioid dependent patients. Drug Alcohol Depend. 2014 Dec 1;145:121-6. doi: 10.1016/j.drugalcdep.2014.10.002. Epub 2014 Oct 16. PMID 25454409
- [Background] Moore MT, Anderson NL, Barnes JM, Haigh EA, Fresco DM. Using the GAD-Q-IV to identify generalized anxiety disorder in psychiatric treatment seeking and primary care medical samples. J Anxiety Disord. 2014 Jan;28(1):25-30. doi: 10.1016/j.janxdis.2013.10.009. Epub 2013 Nov 20. PMID 24334213
- [Background] Newman, M. G., Zuellig, A. R., Kachin, K. E., Constantino, M. J., Przeworski, A., Erickson, T., & Cashman-McGrath, L. (2002). Preliminary reliability and validity of the Generalized Anxiety Disorder Questionnaire-IV: A revised self-report diagnostic measure of generalized anxiety disorder. Behavior Therapy, 33(2), 215-233. https://doi.org/10.1016/S0005-7894(02)80026-0
- [Background] Pani PP, Vacca R, Trogu E, Amato L, Davoli M. Pharmacological treatment for depression during opioid agonist treatment for opioid dependence. Cochrane Database Syst Rev. 2010 Sep 8;(9):CD008373. doi: 10.1002/14651858.CD008373.pub2. PMID 20824876
- [Background] Stathopoulou G, Pollack MH, Otto MW. Anxiety sensitivity moderates drug cravings in response to induced negative affect in opioid dependent outpatients. Addict Behav. 2018 Sep;84:75-78. doi: 10.1016/j.addbeh.2018.03.020. Epub 2018 Mar 13. No abstract available. PMID 29631093
- [Background] Stein MD, Santiago Rivera OJ, Anderson BJ, Bailey GL. Perceived need for depression treatment among persons entering inpatient opioid detoxification. Am J Addict. 2017 Jun;26(4):395-399. doi: 10.1111/ajad.12554. Epub 2017 Apr 28. PMID 28453912
- [Background] Walker J, Burke K, Wanat M, Fisher R, Fielding J, Mulick A, Puntis S, Sharpe J, Esposti MD, Harriss E, Frost C, Sharpe M. The prevalence of depression in general hospital inpatients: a systematic review and meta-analysis of interview-based studies. Psychol Med. 2018 Oct;48(14):2285-2298. doi: 10.1017/S0033291718000624. Epub 2018 Mar 26. PMID 29576041
- [Background] Watkins KE, Hunter SB, Wenzel SL, Tu W, Paddock SM, Griffin A, Ebener P. Prevalence and characteristics of clients with co-occurring disorders in outpatient substance abuse treatment. Am J Drug Alcohol Abuse. 2004 Nov;30(4):749-64. doi: 10.1081/ada-200037538. PMID 15624547
- [Background] Wickersham JA, Azar MM, Cannon CM, Altice FL, Springer SA. Validation of a Brief Measure of Opioid Dependence: The Rapid Opioid Dependence Screen (RODS). J Correct Health Care. 2015 Jan;21(1):12-26. doi: 10.1177/1078345814557513. PMID 25559628
- [Background] Wilhelm S, Weingarden H, Ladis I, Braddick V, Shin J, Jacobson NC. Cognitive-Behavioral Therapy in the Digital Age: Presidential Address. Behav Ther. 2020 Jan;51(1):1-14. doi: 10.1016/j.beth.2019.08.001. Epub 2019 Aug 8. PMID 32005328
- [Background] Gratz, K.L., Roemer, L. Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difficulties in Emotion Regulation Scale. J Psychopathol Behav Assess 30, 315 (2008). https://doi.org/10.1007/s10862-008-9102-4

RESULTS

PARTICIPANT FLOW:
Groups:
- Smartphone Digital Intervention Group: Participants in the smartphone digital intervention group downloaded the "Mood Triggers" application and were asked to engage with the intervention four to six times per week for four weeks, completing 20 brief (~2 minute) CBT-based video sessions. The app passively collected data on ambient light, GPS location, call/text logs, and screen time. Each video guided participants through exercises designed to manage anxiety and depression symptoms, such as progressive muscle relaxation and problem-solving strategies. The videos were categorized into modules including Actions, Mental Hygiene, Exposure, Acceptance, Cognitions, Regulation and Positive Feelings, and Preparation. The app also included optional daily prompts on mood and anxiety, adapted from the PANAS-X, to encourage self-monitoring.
- Wait List Control Condition: The waitlist control group did not receive the digital intervention treatment during the eight-week study. Participants in this group were offered access to the intervention after completing the study. A phone onboarding session was available but not mandatory for the control group, unlike the intervention group.
Period: Overall Study
Arm/Group | Smartphone Digital Intervention Group | Wait List Control Condition
Started | 32 | 31
Completed | 27 | 29
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Smartphone Digital Intervention Group: The Smartphone Digital Intervention Group was the experimental group. Participants randomized to this group downloaded the "Mood Triggers" smartphone application and were asked to use it 4-6 times per week for four weeks, completing 20 digital video sessions. The app passively and continuously collected data on ambient light, GPS location, call and text logs, and screen time. The intervention, based on cognitive-behavioral therapy (CBT) principles, delivered brief informational videos (averaging ~2 minutes) that guided participants through exercises to manage symptoms of anxiety and depression. Examples of these exercises included progressive muscle relaxation, problem-solving strategies, and relapse prevention. The app also featured optional daily prompts, adapted from the PANAS-X, to encourage self-monitoring of mood and anxiety. The videos were organized into modules addressing actions, mental hygiene, exposure, acceptance, cognitions, regulation and positive feelings, and preparation.
- Wait List Control Condition: The waitlist control group did not receive the digital intervention treatment during the eight-week study. They provided urine samples bi-weekly and were offered access to the digital intervention after completing their study participation.
- Total: Total of all reporting groups
Arm/Group | Smartphone Digital Intervention Group | Wait List Control Condition | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.74 (9.20) | 35.47 (9.89) | 37.08 (9.62)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Man | 18 | 14 | 32
  Gender: Woman | 13 | 16 | 29
  Gender: Prefer not to disclose | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 27 | 17 | 44
  Race: Other/multiracial | 4 | 12 | 16
  Race: Prefer not to disclose | 1 | 2 | 3
Depression Severity as Measured by the Patient Health Questionnaire-9 (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report instrument used to assess the severity of depressive symptoms. Each item is scored on a scale from 0 ("not at all") to 3 ("nearly every day"), resulting in a total score range of 0 to 27. Higher scores indicate greater depression severity.
  units on a scale | 16.05 (6.37) | 16.41 (6.04) | 16.23 (6.16)
Anxiety Severity as Measured by the Generalized Anxiety Disorder Questionnaire-IV (GAD-Q-IV) [Mean (Standard Deviation); unit: units on a scale] — The Generalized Anxiety Disorder Questionnaire-IV (GAD-Q-IV) is a 14-item self-report measure used to assess the severity of Generalized Anxiety Disorder (GAD) based on DSM-IV criteria. Possible total scores range from 0 to 12, with higher scores representing greater GAD symptom severity.
  units on a scale | 10.13 (2.17) | 10.18 (2.2) | 10.15 (2.17)
Opioid Use Disorder Severity as Measured by the Rapid Opioid Dependence Screen (RODS) [Mean (Standard Deviation); unit: units on a scale] — Opioid Dependency Using the Rapid Opioid Dependence Screen
  The Rapid Opioid Dependence Screen (RODS) is an 8-item measure assessing opioid dependence. For this study, a total score was calculated by summing two components:
  The number of endorsed opioid types from Item 1 (which lists 8 types, score range 0-8).
  The number of "yes" responses to the 7 dependence-related questions in Items 2-8 (score range 0-7).
  This method results in a total possible score range of 0 to 15. Higher scores indicate both a greater breadth of lifetime opioid use and a higher number of opioid dependence symptoms.
  units on a scale | 8.79 (0.75) | 8.82 (0.62) | 8.80 (0.68)
Opioid Craving Severity as Measured by the Opioid Craving Scale (OCS) [Mean (Standard Deviation); unit: units on a scale] — The Opioid Craving Scale (OCS) is a 3-item self-report measure used to assess opioid craving. Each of the three items is rated on a scale from 0 to 9. The total score is calculated by taking the average of the three item scores, resulting in a final score range of 0 to 9. Higher scores indicate a greater severity of craving.
  units on a scale | 6.54 (3.91) | 6.35 (3.21) | 6.45 (3.56)

OUTCOME MEASURES:

1. Primary Outcome: Change in Anxiety Symptoms as Assessed by Generalized Anxiety Disorder- Q-IV Scale
Description: Assesses anxiety symptoms. Possible GAD-Q-IV scores range from 0 to 12, with higher scores representing greater GAD symptom severity
Time Frame: From Baseline to 4 weeks (post-intervention) and from Baseline to 8 weeks (follow-up).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Smartphone Digital Intervention Group (Experimental Group): Participants in the smartphone digital intervention group downloaded the "Mood Triggers" application and were asked to engage with the intervention four to six times per week for four weeks, completing 20 brief (~2 minute) CBT-based video sessions. The app passively collected data on ambient light, GPS location, call/text logs, and screen time. Each video guided participants through exercises designed to manage anxiety and depression symptoms, such as progressive muscle relaxation and problem-solving strategies. The videos were categorized into modules including Actions, Mental Hygiene, Exposure, Acceptance, Cognitions, Regulation and Positive Feelings, and Preparation. The app also included optional daily prompts on mood and anxiety, adapted from the PANAS-X, to encourage self-monitoring.
Arm/Group | Smartphone Digital Intervention Group (Experimental Group) | Wait List Control Condition
Number analyzed (Participants) | 32 | 31
units on a scale
  Pre-Post | -1.8 [-4.36 to 0.76] | -1.04 [-5.37 to 3.28]
  Pre-Followup | -2.47 [-5.72 to 0.78] | -1.53 [-4.64 to 1.59]
Statistical Analysis 1: Comparison: Smartphone Digital Intervention Group (Experimental Group) vs Wait List Control Condition; Test type: Other; p = .755, Robust linear mixed models; Differences in slopes = 0.76, 95% CI 2-sided [-4.14 to 5.66]

2. Primary Outcome: Change in Depressive Symptoms as Assessed by Patient Health Questionnaire-9
Description: Assesses depressive symptoms, the PHQ-9 score can range from 0 to 27, since each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day)
Time Frame: From Baseline to 4 weeks (post-intervention) and from Baseline to 8 weeks (follow-up).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Smartphone Digital Intervention Group (Experimental Group) | Wait List Control Condition
Number analyzed (Participants) | 32 | 31
units on a scale
  pre-post | -4.03 [-9.07 to 1] | -2.65 [-8.34 to 3.04]
  pre-followup | -5.36 [-11.29 to 0.57] | -1.45 [-5.73 to 2.84]
Statistical Analysis 1: Comparison: Smartphone Digital Intervention Group (Experimental Group) vs Wait List Control Condition; Test type: Other; p = 0.713, Robust linear mixed models; Differences in slopes = 1.38, 95% CI 2-sided [-6.15 to 8.91]

3. Primary Outcome: Change in Likelihood of a Positive Urine Screen for Opioids (MOP)
Description: This outcome measures the change in the likelihood of a positive urine drug screen (UDS) for opioids (MOP). The result of each UDS was coded as a binary variable (0 = negative test, 1 = positive test). The reported data are the beta coefficients (estimated mean change) from a robust linear mixed-effects model, which are presented on a unitless scale. A negative value indicates a reduction in the likelihood of testing positive and represents a better outcome.
Time Frame: From Baseline to 4 weeks (post-intervention) and from Baseline to 8 weeks (follow-up).
Measure: Mean (95% Confidence Interval); unit: beta coefficient
Arm/Group | Smartphone Digital Intervention Group (Experimental Group) | Wait List Control Condition
Number analyzed (Participants) | 32 | 31
beta coefficient
  pre-post | -0.71 [-1.81 to 0.39] | 0.33 [-1.29 to 1.94]
  pre-followup | -0.62 [-1.83 to 0.59] | 1.09 [-0.74 to 2.92]
Statistical Analysis 1: Comparison: Smartphone Digital Intervention Group (Experimental Group) vs Wait List Control Condition; Test type: Other; p = 0.323, Robust linear mixed models; Differences in slopes = 1.03, 95% CI 2-sided [-1.02 to 3.09]

4. Secondary Outcome: Change in Opioid Use Disorder Severity as Measured by the Rapid Opioid Dependence Screen (RODS)
Description: The Rapid Opioid Dependence Screen (RODS) is an 8-item measure used to assess opioid dependence severity. For this study, a total score was calculated by summing two components: 1) The number of endorsed opioid types from Item 1 (which lists 8 types, range 0-8), and 2) The number of "yes" responses to the 7 dependence-related questions in Items 2-8 (range 0-7). This method results in a total possible score range of 0 to 15. Higher scores indicate a greater breadth of lifetime opioid use and a higher number of dependence symptoms. A reduction in score represents improvement.
Time Frame: From Baseline to 4 weeks (post-intervention) and from Baseline to 8 weeks (follow-up).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Smartphone Digital Intervention Group (Experimental Group) | Wait List Control Condition
Number analyzed (Participants) | 32 | 31
units on a scale
  pre-post | -5.23 [-6.37 to -4.1] | -5.56 [-6.96 to -4.15]
  pre-followup | -4.72 [-6.36 to -3.08] | -4.29 [-7.54 to -1.03]
Statistical Analysis 1: Comparison: Smartphone Digital Intervention Group (Experimental Group) vs Wait List Control Condition; Test type: Other; p = .692, Robust linear mixed models; Differences in slopes = -0.33, 95% CI 2-sided [-1.95 to 1.30]

5. Secondary Outcome: Change in Opioid Craving as Measured by the Opioid Craving Scale (OCS)
Description: Opioid Craving Scale (OCS) is a 3-item self-report measure used to assess opioid craving. Each of the three items is rated on a scale from 0 to 9. The total score is calculated by taking the average of the three item scores, resulting in a final score range of 0 to 9. Higher scores indicate a greater severity of craving. A reduction in score represents improvement.
Time Frame: From Baseline to 4 weeks (post-intervention) and from Baseline to 8 weeks (follow-up).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Smartphone Digital Intervention Group (Experimental Group) | Wait List Control Condition
Number analyzed (Participants) | 32 | 31
units on a scale
  pre-post | 0.46 [-1.04 to 1.96] | -1.83 [-4.87 to 1.19]
  pre-followup | 0.06 [-2.25 to 2.36] | -1.61 [-4.38 to 1.16]
Statistical Analysis 1: Comparison: Smartphone Digital Intervention Group (Experimental Group) vs Wait List Control Condition; Test type: Other; p = 0.1, Robust linear mixed models; Differences in slopes = -2.92, 95% CI 2-sided [-6.41 to 0.58]

ADVERSE EVENTS:
Time Frame: From baseline until study completion at 8 weeks.
Description: Adverse events were not systematically collected. Information was collected only when participants voluntarily disclosed adverse events to the study team.
Arm/Group | Smartphone Digital Intervention Group (Experimental Group) | Wait List Control Condition
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT05047627/Prot_SAP_000.pdf